CLINICAL TRIAL: NCT03779750
Title: CausesOf End Stage Renal Disease In Patients Undergoing Regular Hemodialysis In Assiut University Hospital
Brief Title: Causes Of End Stage Renal Disease In Patients Undergoing Regular Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hudna abdullah, Principal Investigator, Assiut University
Other Study IDs: COESRDIPURHIAUH
Record Dates: First submitted 2018-05-20; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: End Stage Renal Disease Patients
MeSH Terms: interventions — Blood Urea Nitrogen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- End Stage Renal Disease Patients: complete blood picture blood urea s.creatinine urine analysis calcium phosphorus parathyroid hormone. 4- Hepatitis BsAg,HCV-Abs and HIV.
  Interventions: Diagnostic Test: s.creatinine

INTERVENTIONS:
Diagnostic Test: s.creatinine — All ESRD patients on regular hemodialysis in dialysis unit of Assiut university Hospital duing one year. will be subjected to 3- Routine investigations including complete blood picture ,blood urea , s.creatinine,urine analysis , calcium, phosphorus, and parathyroid hormone.
  Other Names: blood urea

SUMMARY:
CKD is defined as kidney damage for ≥3 months, as defined by structural and or functional abnormalities of the kidney, with or without decreased GFR or GFR <60 mL/min/1.73m2 for ≥3 months, with or without kidney damage. CKD is classified based on cause, GFR category, and albuminuria category (CGA). ESRD has become a public health problem worldwide, with recent reports showing that the total number of ESRD patients has been growing dramatically.

DETAILED DESCRIPTION:
The prevalence ESRD undergoing maintenance dialysis in 2010 was 284 individuals per million population (pmp) worldwide, which has increased 1.7 times from 165 pmp patients in 1990.

In Egypt, the prevalence of dialysis patients has increased from 225 pmp in 1996 to 483 pmp in 2008(according to last Egyptian renal registry) and the main causes of ESKD in Egypt, other than diabetic nephropathy, included hypertensive kidney disease, chronic glomerulonephritis, unknown etiology, chronic pyelonephritis, schistosomal obstructive uropathy, and schistosomal nephropathy .

It is well established that diabetic kidney disease is the most common cause or in combination with hypertensive nephropathy are the most common causes of end-stage renal disease (ESRD) in developed and developing countries. Patient survival in diabetics on maintenance renal replacement therapy including hemodialysis (HD), peritoneal dialysis (PD) and kidney transplantation is significantly lower than that seen in nondiabetics with ESRD. The poor prognosis of diabetic patients with ESRD is partly due to presence of significant cardiovascular disease, problems with vascular access, more susceptible to infections, foot ulcer, and hemodynamic instability during HD.

Hemodialysis (HD) is the first line of renal replacement therapy in the investigator's country. It is well known that patients on RRT are of greater risk for complications and worse prognosis in comparison to patients with the same co-morbidities but not on RRT.

The most common complicatons of hemodialysis are hypotensive episodes, muscular cramps, itching, arrhythmias,and anaphylactic responses during the sessions.

ELIGIBILITY:
Inclusion Criteria:

* All ESRD patients >18years old in Assuit University Hospital dialysis unit .
* Patients on regular haemodialysis for more than six months.

Exclusion Criteria:

* ESRD patients<18years old .
* patients with acute kidney injury .
* patients on haemodialysis for less than six months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All ESRD patients on regular hemodialysis in dialysis unit of Assiut university Hospital duing one year.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
To find out the possible etiologies of ESRD in patients undergoing regular hemodialysis in Assiut university hospital. | Within one year
  * prevalence of ESRD on regular hemodialysis(in percentage )among different age groups ( measured by years)
  * frequencies(in percentage)of different etiologies in ESRD on regular hemodialysis.
To do registration for ESRD patients undergoing regular haemodialysis in assuit university hospital dialysis unit | Within one year
  • Relation between different causes of ESRD and life expectance.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa A Haridy, Prof.Dr, Principal Investigator — Unaffiliation
Locations (2):
- Egypt (2):
  - Assiut University Hospital, Asyut
  - Hudna Abdullah Ahmed, Asyut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Solomon R. PRESERVE: The End or the Beginning of a New Era in Prevention of Contrast-Associated Acute Kidney Injury? Am J Kidney Dis. 2018 Sep;72(3):322-324. doi: 10.1053/j.ajkd.2018.03.013. Epub 2018 May 8. No abstract available. PMID 29751980
- [Background] Thomas B, Wulf S, Bikbov B, Perico N, Cortinovis M, Courville de Vaccaro K, Flaxman A, Peterson H, Delossantos A, Haring D, Mehrotra R, Himmelfarb J, Remuzzi G, Murray C, Naghavi M. Maintenance Dialysis throughout the World in Years 1990 and 2010. J Am Soc Nephrol. 2015 Nov;26(11):2621-33. doi: 10.1681/ASN.2014101017. Epub 2015 Jul 24. PMID 26209712
- [Background] Ghaderian SB, Hayati F, Shayanpour S, Beladi Mousavi SS. Diabetes and end-stage renal disease; a review article on new concepts. J Renal Inj Prev. 2015 Jun 1;4(2):28-33. doi: 10.12861/jrip.2015.07. eCollection 2015. PMID 26060834
- [Background] Ikizler TA, Schulman G. Hemodialysis: techniques and prescription. Am J Kidney Dis. 2005 Nov;46(5):976-81. doi: 10.1053/j.ajkd.2005.07.037. No abstract available. PMID 16253743